CLINICAL TRIAL: NCT06832787
Title: Prospective, Multi-Center Randomized Controlled Trial for the Combinational Use of Negative Pressure Wound Therapy (NPWT) for the Treatment of Diabetic Wounds
Brief Title: Evaluation of Combinational Use of Negative Pressure Wound Therapy (NPWT) for Diabetic Foot Wounds
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024/2226
Record Dates: First submitted 2025-02-11; First posted 2025-02-18 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-02

CONDITIONS: Diabetic Foot Ulcer
Keywords: Diabetic Foot Ulcer; Negative Pressure Wound Therapy; Dermal Substitute; Delayed wound closure
MeSH Terms: conditions — Diabetic Foot | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NPWT Only (Other): Control: Negative Pressure Wound Therapy only
  Interventions: Device: Negative Pressure Wound Therapy
- NPWT + Kerecis (Active Comparator): Combinational Therapy of Negative Pressure Wound Therapy + application of Kerecis Omega 3 Wound Matrix
  Interventions: Device: Negative Pressure Wound Therapy; Device: Kerecis
- NPWT + Delayed Primary Closure with Local Flap (Active Comparator): Combinational Therapy of Delayed Primary Closure with Local Flap and Negative Pressure Wound Therapy
  Interventions: Device: Negative Pressure Wound Therapy; Device: Delayed primary closure with local flap

INTERVENTIONS:
Device: Negative Pressure Wound Therapy — NPWT applied over wound without any adjuncts
Device: Kerecis — Kerecis Omega3 Wound Dressing is derived from fish skin and is used as a dermal substitute.
  Arms: NPWT + Kerecis
Device: Delayed primary closure with local flap — Delayed primary closure with local flap to close wound
  Arms: NPWT + Delayed Primary Closure with Local Flap

SUMMARY:
Singapore has one of the world's highest diabetes-related lower limb amputation rates in the world. Between 2008 - 2017, 4724/5306 (89.0%) of all major amputations and 6656/7227 (92.1%) of all toe/ray amputations performed in Singapore were for diabetic patients. Diabetic foot ulcers are generally slow to heal and poor wound management may lead to infection and subsequently major amputations. Hence, adequate wound care to achieve wound healing efficiently and effectively is of utmost importance.

In the investigators' clinical practice, Negative Pressure Wound Therapy has been the dressing of choice to aid wound closure and prevent infective complications. Drainage of wound exudates helps to reduce and prevent infection, promote granulation tissue proliferation and induce cell growth. When used in combination with dermal substitutes, graft uptake is improved by further promoting proliferation and encouraging tissue regeneration.

Wounds can also be closed surgically though primary closure, where the skin is closed and serves as a physical barrier against infection. The technique is not without its pros and cons. Primary closure may decrease healing time and reduce need for additional surgery, but these patients are also at risk of recurrent infection and may require more proximal amputation. These may be circumvented with delayed primary closure, which is the surgical closure of the amputation wound at a delayed timing after amputation. This gives the clinical team time to optimize the wound and ensure that there is no underlying infection prior to closure.

The experience of NPWT + Kerecis Omega 3 and delayed primary closure have been positive. To the investigators' current knowledge, there is only one case series reported for the use of fish skin graft in combination with NPWT for the treatment of acute pediatric wounds and two case series for the use of NPWT in diabetic foot wound that has undergone surgical closure. The proposed study would be the first RCT to evaluate effects of combination therapy in both open and closed diabetic foot ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-100
* First or last toe ray amputation
* Adequate perfusion (either >50% stenosis on duplex ultrasound or undergone successful revascularization with <30% residual stenosis)

Exclusion Criteria:

* Amputations not at first or last toe
* Venous ulcers
* Heel ulcers
* Osteomyelitis
* Active Infection
* Patients on imunosuppressant
* Patients with known allergy to fish
* Patients unable to give informed consent.

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-07-22 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of 100% Wound Closure at 12 weeks | 12 weeks post-intervention
  100% Wound Closure defined as re-epithelization without any need for dressing

SECONDARY OUTCOMES:
Time in days taken to achieve complete wound closure | Up to 12 weeks post-intervention
  Time (in days) taken from intervention to 100% wound closure
Change in Wong-Baker FACES® Pain Rating Scale Score from Baseline to 12 weeks | From time of intervention to 12 weeks post-intervention
  Pain score is measured using the Wong-Baker FACES® Pain Rating Scale. Participants will be asked at baseline, and at 4, 8 and 12 weeks subsequently. 0 corresponds to "no pain", and 10 corresponds to "worst pain imaginable".
Occurrence of infection during study period | Up to 12 weeks post-intervention
  Occurrence of any infection at index wound during follow-up period is recorded
Occurrence of further minor amputation during study period | Up to 12 weeks post-intervention
  Occurrence of further minor amputation at index wound during follow-up period is recorded
Occurrence of major amputation during study period | Up to 12 weeks post-intervention
  Occurrence of major amputation at index limb during follow-up period is recorded
Occurrence of death during study period | Up to 12 weeks post-intervention
  Occurrence of death during follow-up period is recorded

CONTACTS AND LOCATIONS:
Overall Officials: Jack Kian Ch'ng, Principal Investigator — Singapore General Hospital
Locations (2):
- Singapore (2):
  - Singapore General Hospital, Singapore
  - Sengkang General Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No
Due to Personal Data Protection Act.

REFERENCES:
- [Background] Ciprandi G, Kjartansson H, Grussu F, Baldursson BT, Frattaroli J, Urbani U, Zama M. Use of acellular intact fish skin grafts in treating acute paediatric wounds during the COVID-19 pandemic: a case series. J Wound Care. 2022 Oct 2;31(10):824-831. doi: 10.12968/jowc.2022.31.10.824. PMID 36240798
- [Background] Aerden D, Vanmierlo B, Denecker N, Brasseur L, Keymeulen B, Van den Brande P. Primary closure with a filleted hallux flap after transmetatarsal amputation of the big toe for osteomyelitis in the diabetic foot: a short series of four cases. Int J Low Extrem Wounds. 2012 Jun;11(2):80-4. doi: 10.1177/1534734612446640. Epub 2012 May 4. PMID 22561521
- [Background] Blume PA, Paragas LK, Sumpio BE, Attinger CE. Single-stage surgical treatment of noninfected diabetic foot ulcers. Plast Reconstr Surg. 2002 Feb;109(2):601-9. doi: 10.1097/00006534-200202000-00029. PMID 11818842
- [Background] Berceli SA, Brown JE, Irwin PB, Ozaki CK. Clinical outcomes after closed, staged, and open forefoot amputations. J Vasc Surg. 2006 Aug;44(2):347-351; discussion 352. doi: 10.1016/j.jvs.2006.04.043. PMID 16890866
- [Background] Zhang L, Weng T, Wu P, Li Q, Han C, Wang X. The Combined Use of Negative-Pressure Wound Therapy and Dermal Substitutes for Tissue Repair and Regeneration. Biomed Res Int. 2020 Dec 4;2020:8824737. doi: 10.1155/2020/8824737. eCollection 2020. PMID 33344649
- [Background] Normandin S, Safran T, Winocour S, Chu CK, Vorstenbosch J, Murphy AM, Davison PG. Negative Pressure Wound Therapy: Mechanism of Action and Clinical Applications. Semin Plast Surg. 2021 Aug;35(3):164-170. doi: 10.1055/s-0041-1731792. Epub 2021 Sep 10. PMID 34526864
- [Background] Riandini T, Pang D, Toh MPHS, Tan CS, Choong AMTL, Lo ZJ, Chandrasekar S, Tai ES, Tan KB, Venkataraman K. National Rates of Lower Extremity Amputation in People With and Without Diabetes in a Multi-Ethnic Asian Population: a Ten Year Study in Singapore. Eur J Vasc Endovasc Surg. 2022 Jan;63(1):147-155. doi: 10.1016/j.ejvs.2021.09.041. Epub 2021 Dec 14. PMID 34916107
- See also: NPWT in closed foot wounds — https://www.researchgate.net/publication/257069667_Use_of_an_Incision-Line_Negative_Pressure_Wound_Therapy_Technique_to_Protect_High-Risk_Diabetic_Foot_Wounds_Postoperatively
- See also: NPWT in closed foot wounds — https://journals.cambridgemedia.com.au/wpr/volume-23-number-1/use-negative-pressure-wound-therapy-dual-closure-and-splinting-device-associated-rapid-delayed-primary-wound-closure-high-risk-d